CLINICAL TRIAL: NCT05913440
Title: A Multicenter Observational Retrospective Study of Therapeutic Approaches and Clinical Outcomes in Real Clinical Practice in Russian Patients With Human Epidermal Growth Factor Receptor 2 (HER2)-Low Unresectable and/or Metastatic Breast Cancer
Brief Title: HER2-low Unresectable and/or Metastatic Breast Cancer in Russia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00029
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Planned study population consists of approximately 3,150 adult patients with HER2-negative (IHC 0, + or IHC2+/ISH-) unresectable or metastatic BC enrolled to the study in order to obtain approximately 2,000 patients with confirmed HER2 low status (IHC1+ or IHC2+/ISH ).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of unresectable and/or metastatic BC established between the 1st July 2021 and the 1st July 2022.
* Patients have HER2-negative status (IHC0, IHC1+, IHC2+/ISH-) obtained in the local laboratory.

  -. Patients have an adequate archival tumor sample and slides suitable for reassessment HER2 status* by the reference laboratory.
* Patients have documented hormonal status (ER, PR) IHC score.
* Age ≥ 18 years at the time of inclusion.
* Patients provided written consent allowing for data and samples to be used in the future and this study would be covered by the consent for future use in accordance with ICH GCP, GPP (Good Pharmacoepidemiology Practices) and local law prior to inclusion in the study. If the patient is deceased, a waiver may be accepted

Exclusion Criteria:

* Patients with previous HER2 positive status in the anamnesis at the diagnosis or after the diagnosis of breast cancer.
* Presence of other malignancies within period since diagnosis until the timepoint of data collection.
* Patients receiving trastuzumab deruxtecan currently or received in anamnesis.
* The participation in any randomised controlled trial within period since diagnosis until end of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Planned study population consists of approximately 3,150 adult patients with HER2-negative (IHC 0, + or IHC2+/ISH-) unresectable or metastatic BC enrolled to the study in order to obtain approximately 2,000 patients with confirmed HER2 low status (IHC1+ or IHC2+/ISH ).
Sampling Method: Non-Probability Sample
Enrollment: 1669 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
To study the overall prevalence of HER2-low among patients with HER2-negative mBC, based on reassessment of historical HER2 fixed tissue IHC stained slides assay in the Russian Federation | 12 months
To study the clinical-pathological, histopathological and demographic profiles of patients of HR-positive and HR-negative HER2-low status among unresectable and/or mBC patients identified as HER2-negative HR-positive/negative | 12 months
  Clinical and demographic data, as well as other study variables will be presented as frequencies or percentages, or as the mean value, standard deviation, median, quantiles, minimum and maximum, depending on the type of variable (continuous or categorical) for the total sample and all subgroups (if applicable).

SECONDARY OUTCOMES:
To describe data on the diagnostic algorithms and therapeutic tactics in patients with HR-positive and HR-negative HER2-low unresectable and/or mBC in routine practice in the Russian Federation | 12 months
  Data on methods used for diagnosis will be presented as frequencies or percentages, or as the mean value, standard deviation, median, quartiles, minimum and maximum, depending on the type of variable (categorical or continuous) for the total sample and all subgroups
To describe data on the treatment approach in patients with HR-positive and HR-negative HER2-low unresectable and/or mBC in routine practice in the Russian Federation, and the sequence of therapy administration (HR-positive and HR-negative). | 12 months
  Data on methods used for anticancer and concomitant treatment will be presented as frequencies or percentages, or as the mean value, standard deviation, median, quartiles, minimum and maximum, depending on the type of variable (categorical or continuous) for the total sample and all subgroups
To assess the treatment outcomes of patients with HR-positive and HR-negative HER2-low unresectable and/or mBC in routine practice in the Russian Federation | 12 months
  Data on methods used for anticancer and concomitant treatment will be presented as frequencies or percentages, or as the mean value, standard deviation, median, quartiles, minimum and maximum, depending on the type of variable (categorical or continuous) for the total sample and all subgroups
To characterize the concordance between HER2 IHC scores in local and reference laboratories after reassessment in the reference lab (IHC 0, 1+, 2+/ISH-) using the existing, and refined, criteria of ASCO/CAP definition | 12 months
  The frequency of concordance of IHC HER2 scores and ISH results between local and reference laboratories will be calculated along with exact 95% CIs. Cohen's Kappa statistics will be used to evaluate concordance between HER2 IHC scores in local and reference laboratories.
To describe the concordance of HER2 status evaluations performed in a reference laboratory by a pathologist manually and by an artificial intelligence (AI) program. | 12 months
  Concordance assessed using Cohen's Kappa statistics (positive, negative and overall agreement) between HER2 status evaluations performed in a reference laboratory by a pathologist manually and by an AI program.

CONTACTS AND LOCATIONS:
Locations (40):
- Russia (40):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Chita
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Istra
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Kemerovo
  - Research Site, Khanty-Mansiysk
  - Research Site, Kirov
  - Research Site, Kostroma
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Maykop
  - Research Site, Moscow
  - Research Site, Nal'chik
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saransk
  - Research Site, Sevedorvinsk
  - Research Site, Smolensk
  - Research Site, Sochi
  - Research Site, Surgut
  - Research Site, Tomsk
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/